CLINICAL TRIAL: NCT02888652
Title: Multivariate Analysis of Platelet Reactivity Variety in Patients With Coronary Heart Disease After PCI
Brief Title: Study on the Registration of Coronary Heart Disease Patients Undergoing PCI
Status: Completed | Type: Observational
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: XY3-CLOP1507A01; ChiCTR-OOC-16009006 (Registry Identifier: Chinese Clinical Trial Registry)
Record Dates: First submitted 2016-08-11; First posted 2016-09-05 (Estimated); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Coronary Heart Disease
Keywords: Coronary Heart Disease; PCI; Anti-Platelet Agents
MeSH Terms: conditions — Coronary Disease | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — gene test
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: antiplatelet agents(Clopidogrel or Ticagrelor) — Clinical physicians according to patients condition to give different antiplatelet agents(Clopidogrel or Ticagrelor).We only observe clinical curative effect.
  Other Names: Clopidogrel or Ticagrelor

SUMMARY:
Study on the registration of coronary heart disease patients undergoing PCI in Chinese's population. Get the incidence of adverse events in these patients after PCI, a clear type of adverse reaction, forms, influencing factors, to establish risk management processes, clinical safety and reasonable treatment, and provide the basis for further research and reference.

DETAILED DESCRIPTION:
Dual antiplatelet therapy, comprising a low-dose aspirin and a kind of P2Y12 Receptor Inhibitors, has been the mainstay of the management in patients with acute coronary syndromes and/or undergoing Percutaneous Coronary Intervention (PCI). While variability to P2Y12 receptor inhibitors is common in patients and is a major cause of adverse cardiovascular events. Low response to P2Y12 receptor inhibitors will result high platelet reactivity (HPR) and patients who exhibit HPR are at increased risk of atherothrombotic occlusion events. Vice versa, high response to P2Y12 receptor inhibitors will lead to low platelet reactivity (LPR) and increase the risk of hemorrhage.Now, the absence of a universal definition of therapeutic window for different racial and actual clinical situations and lacking the gold standard test to quantify it limit the use in clinic practice.So this clinical trial try to use patient's platelet reactivity combine with type of adverse reaction, forms, influencing factors to find a proper therapeutic windows for P2Y12 receptor inhibitors in Chinese people.

ELIGIBILITY:
Inclusion Criteria:

* Chinese's patients diagnosed with coronary heart disease and accept stent implantation.
* Accept aspirin and P2Y12 receptor inhibitors (clopidogrel or ticagrelorwere）after stent implantation.
* Willingness and ability to sign informed consent.
* Can communicate effectively and complete the trial.

Exclusion Criteria:

* Occurrence of a major complication during the procedure of percutaneous coronary intervention or before platelet function testing.
* Allergy or intolerance to aspirin or P2Y12 receptor inhibitors (Clopidogrel or Ticagrelor）

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with coronary artery disease treated with aspirin and clopidogrel after successful stent implantation.
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | within 1 year after PCI
  ischemic and bleeding

SECONDARY OUTCOMES:
Blood drug concentration | at 5-7 days, 1month, 3 months, 6 months and 12 months after taking anti-platelet agents
  Clopidogrel and Ticagrelor
Mild to moderate adverse events | within 1 year after PCI
  renal function
Platelet activity | at 12- 24 hours, 1 month, 3 months, 6 months and 12 months after PCI
  Platelet activity

CONTACTS AND LOCATIONS:
Overall Officials: GuoPing Yang, professor, Principal Investigator — The Third Xiangya Hospital of Central South University; Yu Cao, MD, Principal Investigator — The Third Xiangya Hospital of Central South University; Jingle Li, MD, Principal Investigator — The Third Xiangya Hospital of Central South University
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China